CLINICAL TRIAL: NCT02134899
Title: An Open-labelled Multicenter Randomized Study on the Efficacy of Everolimus in Reducing Total Native Kidney Volume in Kidney Transplanted Patients With Autosomal Dominant Polycystic Kidney Disease
Brief Title: The Efficacy of Everolimus in Reducing Total Native Kidney Volume in Polycystic Kidney Disease Transplanted Recipients
Acronym: EVERKYSTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P 090804; 2012-004265-41 (EudraCT Number)
Record Dates: First submitted 2014-04-28; First posted 2014-05-09 (Estimated); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Autosomal dominant polycystic kidney disease; cyst; kidney; liver; kidney transplantation; IF/TA; fibrosis; DSA; mTOR inhibitors; calcineurin inhibitors
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Cysts; Fibrosis | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Everolimus (Experimental): everolimus based immunosuppression
  Interventions: Drug: Everolimus
- Calcineurin (Active Comparator): Calcineurin inhibitors maintenance
  Interventions: Drug: Calcineurin inhibitors maintenance

INTERVENTIONS:
Drug: Everolimus — Change from a calcineurin inhibitors-based immunosuppression to an everolimus-based immunosuppression
  Other Names: everolimus conversion
  Arms: Everolimus
Drug: Calcineurin inhibitors maintenance — Usual treatment
  Other Names: calcineurin-inhibitors based immunosuppression
  Arms: Calcineurin

SUMMARY:
The investigators multicenter randomized open-labelled study will investigate the efficacy of an everolimus based immunosuppression in reducing total native kidney volume in kidney recipients with autosomal dominant polycystic kidney disease compared to a calcineurin inhibitor-based immunosuppression.

DETAILED DESCRIPTION:
Kidney graft recipients receiving a firs kidney graft (between 6 months and 5 years post-transplantation) will be randomized 1:1 to receive an everolimus based immunosuppression (in association with steroids and mycophenolate mofetil) or to continue their calcineurin inhibitor-based immunosuppression regimen. The primary objective will be the reduction of total native kidney volume after a 2-years treatment period.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years-old
* recipients of a first kidney graft between 6 month and 5 years ago with a stable eGFR above 30 ml/min/1,73m2
* contraception for female recipients to avoid pregnancy
* valid health Insurance during the study period

Exclusion Criteria:

* signed informed consent not obtained

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-10-14 (Actual); Primary Completion 2017-11-11 (Actual); Study Completion 2017-11-11 (Actual)

PRIMARY OUTCOMES:
Total native kidney volume variation | 24 months after randomization
  measurements of total native kidney volume with a MRI

SECONDARY OUTCOMES:
Volume variation of the biggest liver cyst | 24 months after randomization
  Measurements of the biggest liver cyst volume with a MRI
Interstitial Fibrosis/Tubular Atrophy variation | 24 months after randomization
  IF/TA quantification using Banff criteria during a kidney biopsy
% interstitial fibrosis using Red Sirius staining | 24 months after randomization
  % fibrosis quantified using a morphometry software
Calculated Estimated Glomerular Filtration rate | At baseline, 1 month, 6 months, 12 months, 18 and 24 months
  calculated estimated GFR
Measured Glomerular Filtration rate | At baseline and 24 months
  measured GFR
Proteinuria | At baseline, 1 month, 6 months, 12 months, 18 and 24 months
  Measurement
systolic and diastolic blood pressure | At baseline, 1 month, 6 months, 12 months, 18 and 24 months
  Clinic measurement
Occurrence of diabetes or hyperlipidemia | up to 24 months
  Measurements
Occurrence of neoplasia | up to 24 months
  Medical chart reporting
Development of HLA Donor Specific Antibody (DSA) | At baseline, 1 month, 6 months, 12 months, 18 and 24 months
  V0, 1 year and 2 years after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Hélène François, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bicêtre Hospital, Le Kremlin-Bicêtre, France